CLINICAL TRIAL: NCT01168765
Title: Tu Salud Si Cuenta: UT Community Outreach Program for Community-based Diabetes Prevention and Control
Acronym: UTCO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Belinda Reininger, Associate Professor, Health Promotion and Behavioral Sciences, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSC-SPH-10-0015; 2010-033710 (Other Grant/Funding Number: Texas Department of State Health Services)
Record Dates: First submitted 2010-07-21; First posted 2010-07-23 (Estimated); Last update posted 2013-05-09 (Estimated); Status verified 2013-05

CONDITIONS: Diabetes, Obesity
Keywords: Physical Activity, Mexican-American, Obesity, Diabetes, Nutrition, Border Health
MeSH Terms: conditions — Diabetes Mellitus; Obesity; Motor Activity | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): This is the promotora plus group that will receive the TSSC newsletter and exposure to the media campaign but will also receive monthly visits by promotoras/lay health workers who will review the monthly newsletter with participants, emphasize role model stories, and discuss physical activity and healthful food choices using motivational interviewing strategies.
  Interventions: Behavioral: Tu Salud Si Cuenta Behavioral Intervention
- Control group (Other): TSSC Media Campaign only participants who will receive a newsletter and the same exposure to the media campaign intervention as other community members not enrolled in the behavioral intervention.
  Interventions: Behavioral: Tu Salud Si Cuenta Behavioral Intervention

INTERVENTIONS:
Behavioral: Tu Salud Si Cuenta Behavioral Intervention — A behavioral intervention to assess the impact of the TSSC Media Campaign intervention outreach components with two study arms. The first arm is comprised of participants enrolled in the TSSC Media Campaign(control group) and the second arm(intervention group)consisting of participants exposed to media campaign who will be exposed to additional outreach efforts by monthly visits from lay health workers.
  Other Names: TSSC Media Campaign Plus Refined Promotora Outreach group.(intervention group); TSSC Media Campaign ONLY group. (Control group)

SUMMARY:
Building from existing intervention strategies designed for the Mexican American population entitled Tu Salud Si Cuenta(TSSC) or Your Health Matters. This intervention highlights in the media successful role models who have changed their food choices and physical activity levels. In addition, the intervention designs environmental changes to help community members carry out recommended behavior change strategies. The purpose of this study is to test the efficacy of the outreach elements of the Tu Salud Si Cuenta (TSSC) media campaign, a physical activity and healthful food choice intervention among Mexican Americans in the Lower Rio Grande Valley to achieve behavioral and clinical outcomes.

DETAILED DESCRIPTION:
The proposed intervention research study is building from existing intervention strategies designed for the Mexican American population entitled Tu Salud Si Cuenta (TSSC) or Your Health Matters. This intervention highlights in the media successful role models who have changed their food choices and physical activity levels. In addition the intervention designs environmental changes to help community members carry out recommended behavior change strategies. Outcomes of interest for this study include increased physical activity so as to achieve the CDC/ACSM recommendations of 150 minutes of moderate to vigorous physical activity each week (Haskell et al., 2007), eating 5 servings of fruits and vegetables each day, reducing food portion sizes, and subsequent changes in biomarkers of health.

To test the efficacy of the outreach components of this campaign we are proposing a behavioral intervention trial with two study arms: 1) media campaign or 2) media campaign plus promotora outreach. Data will be collected from the 500 newly enrolled members of the Cameron County Hispanic Cohort, each member from a different household and primarily from quartiles two and four. The measures of this group will be the standard measures collected from the cohort including their medical history, clinical measures and behavioral measures. Two additional measures specified in this proposal will be obtained.

Participants assigned to the TSSC media campaign-only arm of the study will receive a welcome TSSC newsletter upon enrollment to the study, and will receive the same exposure to the TSSC media campaign as other community members not enrolled in the behavioral intervention trial. This includes exposure to the campaign when at the Clinical Research Unit for CCHC data collection via possible viewing of TSSC television segments in the waiting area, and availability of TSSC newsletters. Other possible TSSC campaign exposure will occur as it does for the general public via radio, television and website, using the walking trials, going to farmers market, etc.

Participants assigned to the Promotora plus arm of the study will also receive the initial welcome TSSC newsletter, and other media campaign materials to assure that they are aware of the various media outlets and programming of the campaign. In addition, they will receive a promotora home visit within two weeks of their enrollment. The home visit will consist of the promotora delivering that month's TSSC newsletter, reviewing the newsletter with the participant, emphasizing the role model story, discussing physical activity and healthful food choices using motivational interviewing strategies. These strategies allow the community member to discuss their own goals for making change on these issues while the promotora reflectively listens and summarizes their comments. During the home visit, the promotora will also invite the participant to relevant and accessible opportunities for physical activity and healthful food choices, such as neighborhood walking groups, exercise classes, Farmers' Market, nutrition and cooking classes. Subsequently a monthly home visit will be made by a promotora to deliver the TSSC newsletter, and to follow-up on the initial conversation and referrals. Monthly visits will be made to all 250 participants in the promotora plus arm of the study. Other tools and resources the promotoras might use at the home visits might include showing the participant how to access recipes and resources on the TSSC website, viewing relevant TSSC TV clips on a laptop. Participants will also be invited to an annual celebration of the TSSC media campaign which will feature speakers, cooking and exercise demonstrations and opportunities for networking.

The purpose of this study is to test the efficacy of the outreach elements of the Tu Salud Si Cuenta (TSSC) media campaign, a physical activity and healthful food choice intervention among Mexican Americans in Lower Rio Grande Valley, to achieve behavioral and clinical outcomes.

Information will be collected from the participants and will be followed every five years under their current cohort protocol.

Data of additional behavioral and clinical measures from these participants will be taken annually for up to five years following the same protocol as used for all CCHC participants and specifically collecting the measures below.

All participants are invited to the Clinical Research Center for Clinical and Translational Sciences (CRC-CTSA) or if they prefer, visited in their home. Following a 10 hour fast, 2 EDTA vials (20 cc) of blood will be collected from a peripheral vein (antecubital fossa). Participants are offered a small snack. Blood samples are placed on ice immediately and processed for cholesterol and triglyceride levels using Cardiochek bioscanners and test strips (Polymer Technology Systems, Inc. Indianapolis, IN). Plasma glucose is measured using a YSI 2300 STAT PLUS-D instrument (YSI, Inc. Yellow Springs, OA). Complete blood count with differential white blood counts is performed on whole blood using a Beckman coulter Ac-T diff analyzer (Beckman-Coulter, Inc. Fullerton, CA). Both EDTA tubes are centrifuged at 4.0 C in a refrigerated centrifuge at 4oC (Labnet International, Inc. Edison, NJ) at 1200 relative centrifugal force for 12 minutes. Plasma is separated, aliquoted and immediately frozen at -70° in more than one freezer at UTSPH-B field research laboratory.

Total cholesterol and triglycerides and lipid profiles are assayed. High Density Lipoprotein (HDL) cholesterol is determined using the precipitation method. Low Density Lipoprotein (LDL) cholesterol is calculated by the Friedewald equation modified to use the factor of triglycerides/5 for adults. In all cases LDL is estimated if triglycerides are less than or equal to 400 mg/dl. Insulin is measured using radioimmunoassay (Diagnostic Products, Inc., Los Angeles, CA) and insulin resistance is calculated using the HOMA equation.

Total glycosylated hemoglobin and Hemoglobin A1c are measured using the principle of boronate affinity and high-performance liquid chromatography (HPLC) and be performed by the clinical laboratory of the Valley Baptist Medical Center (Harlingen, TX). C-reactive protein (CRP) is measured at the UTSPH-B field research laboratory using ELISA (Alpha Diagnostics Intl. Inc. San Antonio, TX) with external quality control performed on randomly selected samples at the Section of Atherosclerosis and Lipoprotein Research located in Baylor College of Medicine (Houston, TX). IL6 and TNFα will be performed using Elisa at the UTSPH-B field research laboratory (BD Biosciences, San Jose, CA).

Survey information is collected from the participants in an interview format during their clinical visit as well. These surveys are conducted throughout the visit to ensure that the CCHC participant time is used wisely. All persons collecting the survey information are trained and monitored. Behavioral and awareness measures are collected. Clinical measures collected from the CCHC participants will be used in this proposed study as well.

All individuals are given an exit interview to review immediate findings. Participants are provided with a written summary including their height, weight, waist circumference, blood pressure, fasting glucose, cholesterol and triglycerides. Values out of their expected range are flagged and referrals made as necessary. This interview is also used to address any questions or concerns that may be raised and uses motivational interview strategies to discuss goal setting.

In addition to the information regularly collected during an enrollment visit to the Cameron County Hispanic Cohort, participants consented for this study will also be asked to complete two additional questionnaires: Diabetes Knowledge and Health Care Utilization

Course of Study: The study will take place for up to 5 years. Participants will be approached for participation in this study as they come for their scheduled visit to the Clinical Research Unit in Brownsville. They will be newly enrolled members of the cohort. Cohort participants are enrolled by selecting random census tracts and random census blocks. All households in the selected census block are eligible to participate in this study but, to avoid clustering within the same household, we plan to select only one household member between age 18-75 to participate in this study. This creates a model where neighbors are enrolled in the cohort. This also allows for neighborhood-based (census block) intervention programming to be conducted by the promotoras. We will be offering referrals to our TSSC exercise groups and walking groups located in the TSSC plus intervention arm blocks as well as regular visits by the promotoras to discuss media and newsletters using Motivational Interviewing Strategies.

ELIGIBILITY:
Inclusion Criteria:

* Mexican American men and women aged between 18-75 years old are eligible. All participants of the Behavioral Intervention Trial will first be newly enrolled participants in the Cameron County Hispanic Cohort(CCHC). Persons involved in other intervention studies are eligible to be included in this study as well.

Exclusion Criteria:

* Mexican American men and women older than 75 years or younger than 18 years will be excluded. Persons not enrolled in CCHC will be excluded.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2010-06; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Outcome of Physical Activity | minutes of physical activity obtained in last 7 days
  Minutes of physical activity obtained during last 7 days and examined annually by study groups over time.
Outcome of Fruit and Vegetable intake | servings of fruits & vegetables consumed daily
  serving of fruits and vegetables consumed daily as determined by pictures of serving sizes and examined annually
Biomarkers | assessed annually by study groups over time
  Biomarkers measured by standardized clinical measurement, as in blood pressure, fasting blood glucose, etc., and assessed annually.

SECONDARY OUTCOMES:
Diabetes knowledge | assessed annually by a measured score on diabetes knowledge survey
  A diabetes knowledge survey will be administered annually and the measurement will be based on the resulting score.
Quality adjusted life years | assessed annually at examination
  Measured according to a score on five constructs(mobility, self-care, usual activities, pain/discomfort, anxiety/depression) and assessed annually.

CONTACTS AND LOCATIONS:
Overall Officials: Belinda Reininger, DrPH, Principal Investigator — University of Texas Health Science Center at Houston School of Public Health-Brownsville Regional Campus
Locations (1):
- University of Texas School of Public Health-Brownsville Regional Campus, Brownsville, Texas, United States

REFERENCES:
- [Derived] Heredia NI, Xu T, Lee M, McNeill LH, Reininger BM. The Neighborhood Environment and Hispanic/Latino Health. Am J Health Promot. 2022 Jan;36(1):38-45. doi: 10.1177/08901171211022677. Epub 2021 Jun 15. PMID 34128383
- [Derived] Vidoni ML, Lee M, Mitchell-Bennett L, Reininger BM. Home Visit Intervention Promotes Lifestyle Changes: Results of an RCT in Mexican Americans. Am J Prev Med. 2019 Nov;57(5):611-620. doi: 10.1016/j.amepre.2019.06.020. Epub 2019 Sep 27. PMID 31564601